CLINICAL TRIAL: NCT06857877
Title: Arlington Study of Healthy Aging
Brief Title: Arlington Aging Study
Status: Recruiting | Type: Observational
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Michael Nelson, Associate Professor, The University of Texas at Arlington
Other Study IDs: 2024-0111
Record Dates: First submitted 2024-09-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Aging
Keywords: Aging; MRI; Cognitive Function; Exercise Science; Remote Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be stored in special tubes that preserve genetic material. Genetic testing experiments, including targeted single variants, single gene testing, genetic panel testing, whole genome sequencing, chromosomal testing, gene expression and biochemical testing, may be performed on the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older Adults

SUMMARY:
The goal of this observational study is to learn about the mechanisms causing functional decline with age, using exercise science, neuroscience, and remote monitoring.

Specific aims include:

Aim 1: Advance knowledge of the biology of aging and its impact on the prevention, progression, and prognosis of disease and disability.

Aim 2: Determine the effects of personal and societal factors on aging.

Aim 3: Examine the influence of racial/ethnic and sex differences on the biology of aging and its impact on the prevention, progression, and prognosis of disease and disability.

DETAILED DESCRIPTION:
Subjects will be asked to participate in two study visits that may last up to 5 hours each. In some cases, additional visits may be needed to accommodate their schedule, and/or the schedule of the study team. All participants will provide informed consent prior to participating in the study procedures such as demographic, medical history, risk factor assessment; questionnaires; geographic information system analysis; blood pressure measurements; assessment of aerobic exercise capacity, cognitive function; olfactory testing; Dual X-Ray absorbency, fasting followed by venous blood draw, vascular function assessment; testing of muscle strength; short physical performance battery; functional mobility; and remote monitoring. The order of procedures and visits may change depending on participant, staff, equipment, and infrastructure availability/needs. Moreover, procedures may be repeated for data quality purposes, if deemed necessary by the investigators.

ELIGIBILITY:
Inclusion Criteria:

Phase 1: Young healthy men and women between 18 - 30 years of age, and older men and women between 50 - 80 years of age.

Phase 2: Men and women living in Tarrant County, Texas, between 50 - 80 years of age. In addition, the investigators will study up to 120 younger men and women, between 18-30 years of age, equally divided by race/ethnicity (same as above) and sex, to serve as reference controls.

Exclusion Criteria:

Phase 1: Clinical diagnosis of dementia; major depression (diagnosed by a physician), visual or auditory impairments that preclude neuropsychological testing or otherwise jeopardize the health and wellbeing of the participant during testing, non-ambulatory status (i.e. less than 10 m without mobility aid), shortness of breath while performing normal activities of daily living (walking through grocery store), body mass index > 45 kg/m2, heart failure or cardiomyopathy, acute coronary syndrome, primary valvular heart disease, severe gait disorder due to musculoskeletal disease or neurological motor deficit (e.g. severe osteoarthritis, lower limb amputation, Parkinson's disease, major stroke with motor sequelae), the use of neuroleptics, participation in a dedicated weight loss program within 6 months before the study; daily consumption of more than two alcoholic beverages; current treatment for cancer, and estimated life expectancy <4 years. Inclusion/exclusion will be verified using the demographics and medical history.

Phase 2: Clinical diagnosis of dementia; major depression (diagnosed by a physician), visual or auditory impairments that preclude neuropsychological testing or otherwise jeopardize the health and wellbeing of the participant during testing, non-ambulatory status (i.e. less than 10 m without mobility aid), shortness of breath while performing normal activities of daily living (walking through grocery store), body mass index > 45 kg/m2, heart failure or cardiomyopathy, acute coronary syndrome, primary valvular heart disease, severe gait disorder due to musculoskeletal disease or neurological motor deficit (e.g. severe osteoarthritis, lower limb amputation, Parkinson's disease, major stroke with motor sequelae), the use of neuroleptics, participation in a dedicated weight loss program within 6 months before the study; daily consumption of more than two alcoholic beverages; current treatment for cancer, and estimated life expectancy <4 years. Inclusion/exclusion will be verified using the demographics and medical history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women currently living in Tarrant County will be contacted through IRB approved flyers, targeted ads (social media), and/or word-of-mouth.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Sense of Smell | Baseline
  Olfactory Testing will be assessed using the NIH Toolbox Odor Identification cards. After scratching a card and sniffing from each sample, respondents will be asked to choose the best match for each odor from pictures representing the odor sources.
Blood Pressure | Baseline
  Blood Pressure will be measured in the sitting position using an automated blood pressure monitor. After sitting blood pressure measurements, participants will be asked to stand up to measure standing blood pressure.
Street Address | Baseline
  Geographic information systems will assign a geocode to each participant's home address, providing latitude, and longitude coordinates based on the provided street address.
Ankle Brachial Index | Baseline
  The Ankle Brachial Index will be noninvasively assessed using the Smartdop XT device (Koven Technology, Inc.).
Pulse Wave Velocity | Baseline
  Arterial stiffness will be measured non-invasively with the Sphygmocor XCEL device (AtCor Medical).
Flow- mediated dilation | Baseline
  The flow-mediated change in brachial artery diameter (i.e. flow-mediated dilation; FMD), in response to a 5-minute period of arterial occlusion will be used to assess peripheral vascular function.
Steps taken | Baseline
  A wrist-worn continuous activity tracker (Fitbit wristband) will be worn by the subjects for 7 days.
Sedentary Time | Baseline
  A wrist-worn continuous activity tracker with heart rate monitor (Fitbit wristband) will be worn by the subjects for 7 days.
Sleep | Baseline
  A wrist-worn continuous activity tracker (Fitbit) will be worn by the subjects for 7 days to assess total sleep time, and sleep quality.
Medical History Questionnaire | Baseline
  Participants will complete health history questionnaires to gain a deeper understanding of their lived experiences and past medical history.
Complete blood count | Baseline
  Venous blood will be drawn by a trained phlebotomist and/or nurse in the fasting state. Blood will be shipped to LabCorp for processing of the complete blood count.
Functional Mobility | Baseline
  Objective gait measurements will be obtained using a gait mat. Participants will complete 6 separate walks down the full length of the walkway; 3 walks at a preferred pace and 3 walks while performing different secondary tasks (i.e. dual-task gait) in a fixed order:
  1. counting backward by ones,
  2. naming animals, and
  3. counting backward by sevens.
  Walking aids will be permitted.
Cognitive Function | Baseline
  Cognitive function will be assessed using the NIH Toolbox Cognition Battery (NIHTB-CB), administered on an iPad or computer by a trained study team member.
Lower extremity function | Baseline
  Participants will perform the Short Physical Performance Battery (SPPB). The test includes walking, the sit-to-stand test and balance.
Grip strength | Baseline
  Grip strength will be measured following a standardized approach using a validated Jamar handgrip dynamometer (Model J00105, JAMAR Hydraulic Hand Dynamometer).
Bone Density | Baseline
  Participants will undergo Dual X-Ray Absorbency (DEXA) to measure bone density.
Interstitial glucose | Baseline
  A continuous glucose monitor that measures interstitial glucose will be worn by the subject for 7 days.
Body Composition | Baseline
  Participants will undergo Dual X-Ray Absorbency (DEXA) to measure subcutaneous and visceral fat content.
Ambulatory blood pressure | Baseline
  A wrist worn continuous blood pressure monitor (Aktiia wristband) will be worn by the subjects for 7 days for the measurement of ambulatory blood pressure.
Exercise Capacity | Baseline
  Exercise Capacity will be assessed using the six-minute walk test.
Blood lipids | Baseline
  Venous blood will be drawn and shipped to Labcorp for blood lipid analysis
Metabolic Panel (blood) | Baseline
  Venous blood will be drawn and shipped to labcorp for evaluation of the metabolic panel.
Apolipoprotein A | Baseline
  Measured by labcrop from venous blood draw.
Apolipoprotein B | Baseline
  Analyzed by labcorp from venous blood draw.
Lipoprotein A | Baseline
  Analyzed by labcorp from venous blood draw
Blood checmistry panel | Baseline
  Analyzed by labcorp from venous blood draw
HbA1C (blood) | Baseline
  Analyzed by labcorp from venous blood draw
High sensitivity C reactive protein (blood) | Baseline
  Analyzed by labcorp from venous blood draw
Genetic testing | Baseline
  Whole blood (approximately 25 ml) will be stored in special tubes that preserve genetic material in our -80ºC freezer. Genetic testing experiments, including targeted single variants, single gene testing, genetic panel testing, whole genome sequencing, chromosomal testing, gene expression and biochemical testing, may be performed on the samples.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided